CLINICAL TRIAL: NCT06159023
Title: Bronchoalveolar Lavage Using a Conventional Bronchoscope vs. Bronchial Washing Using a Thin Bronchoscope to Diagnose Pulmonary Tuberculosis: a Prospective Randomized Trial
Brief Title: Conventional Bronchoscope With BAL vs. Thin Bronchoscope With BW to Diagnose Pulmonary TB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TBBR trial
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thick scope + BAL (No Intervention): In this arm, participants with suspected pulmonary TB will be received bronchoscopic procedure using thick (5.9mm diameter) conventional bronchoscope and bronchoalveolar lavage (BAL).
- Thin scope + BW (Experimental): In this arm, participants with suspected pulmonary TB will be received bronchoscopic procedure using thin (4.0mm diameter) bronchoscope and bronchial washing (BW).
  Interventions: Device: bronchial washing using a thin bronchoscope

INTERVENTIONS:
Device: bronchial washing using a thin bronchoscope — For intervention, we plan to perform bronchial washing using a thin bronchoscope instead of bronchoalveolar lavage with the conventional thick bronchoscope to diagnose pulmonary TB.
  Arms: Thin scope + BW

SUMMARY:
This study aims to compare the diagnostic yield of bronchoalveolar lavage (BAL) using a thick conventional bronchoscope and bronchial washing (BW) using a thin bronchoscope in the diagnosis of pulmonary tuberculosis.

DETAILED DESCRIPTION:
In patients with suspected pulmonary tuberculosis (TB), confirm the presence of TB bacilli through sputum testing is essential for diagnosis. However, the sensitivity of sputum specimens is suboptimal, and some patients may be unable to produce sputum. In such situations, it is traditionally known that obtaining samples through bronchoscopy increases the diagnostic yield of pulmonary TB. Typically, the method of using a thick, conventional bronchoscope to perform bronchial washing (BW) or bronchoalveolar lavage (BAL) is commonly employed. However, a drawback of the conventional bronchoscope is its inability to reach close to peripheral pulmonary TB lesions due to its larger diameter.

Recent studies have reported an increased diagnostic yield for pulmonary TB when using a thin bronchoscope for BW compared to using a thick, conventional bronchoscope for BW. However, a direct comparison with the method of performing BAL (BAL may have a higher diagnostic yield compared to BW) using a conventional bronchoscope has not been conducted. This study aims to prospectively compare the diagnostic yield for pulmonary TB between BAL using a conventional bronchoscope and BW using a thin bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

* participants age > 17 years with suspected pulmonary TB
* possible active pulmonary TB evident on chest radiography or CT scan
* negative AFB smear results (using two consecutive self-expectorated sputum)
* negative TB-PCR results (using one self-expectorated sputum)
* inability to produce self-expectorated sputum

Exclusion Criteria:

* a request for empirical TB treatment rather than bronchoscopy
* suspect pulmonary TB lesions that are difficult to target for BAL or BW (e.g., multiple discrete tiny nodules)
* contra-indication of bronchoscopy (e.g., bleeding tendency, hypoxemia requiring oxygen, or uncontrolled cardio/cerebrovascular disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TB detection rate | within 2 weeks of bronchoscopy
  Positivity rate of Xpert MTB/RIF assay in BAL or BW fluid

SECONDARY OUTCOMES:
Mycobacterium tuberculosis culture | within 8 weeks of bronchoscopy
  Positivity rate of Mycobacterium tuberculosis culture in BAL or BW fluid
AFB(acid-fast bacilli) smear | within 2 weeks of bronchoscopy
  Positivity rate of AFB smear in BAL or BW fluid
Adverse event | within 2 weeks of bronchoscopy
  Adverse event related/unrelated to bronchoscopy
Time to treatment | within 8 weeks of bronchoscopy
  Time to treatment (TB treatment commencing date - bronchoscopy date, day) in participants with confirmed TB

CONTACTS AND LOCATIONS:
Overall Officials: Jeongha Mok, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No